CLINICAL TRIAL: NCT02778646
Title: Detection of Familial Hypercholesterolaemia Within United Kingdom Based National Disease Registries: A National Institute for Cardiovascular Outcomes Research (NICOR) Study
Brief Title: Detection of Familial Hypercholesterolaemia in Cardiovascular Disease Registry
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NCR-15-07
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2015-07

CONDITIONS: Familial Hypercholesterolemia; Cardiac Event; Percutaneous Coronary Intervention
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

GROUPS / COHORTS (2):
- MINAP Audit: Individuals within this group are those that have been admitted into a United Kingdom (UK) based hospital following a major cardiac event. The FH status of individuals within this group is unknown.
- BCIS Audit: Individuals within this group are those who have undergone percutaneous coronary intervention in the United Kingdom (UK). The FH status of individuals within this group is unknown.

SUMMARY:
Familial hypercholesterolaemia (FH) is an autosomal dominant somatic mutation commonly located on the LDL-receptor, APOB, and PCKS9 gene. The estimated prevalence of homozygous FH is estimated at 1 in a million, whereas the prevalence of heterozygous FH ranges from 1/500-1/200 (0.2-0.5%) of the general population. The majority of individuals suffering from FH remain undiagnosed and without treatment. Using preexisting clinical guidelines, this study scored patients within national cardiovascular disease (CVD) registries for FH with the aim of evaluating prevalence of FH among individuals suffering from premature cardiac events within the UK.

Following scoring of the registry, this study also examined the relationship between cholesterol and survival after a premature event in order to understand the possible ramifications of untreated FH on patient survival.

DETAILED DESCRIPTION:
Familial Hypercholesterolaemia (FH) is a genetic disorder caused by a mutation in the low-density lipoprotein receptor (LDL-R) gene. Individuals suffering from FH experience elevated cholesterol levels that are outside of the accepted range of healthy cholesterol levels. When left untreated FH may cause complications in cardiovascular health and may cause premature cardiac events. Current screening methods for this disease do not successfully diagnose the majority of FH cases.

This study applies three clinical diagnostic tools--Dutch Lipid Clinic Network Criteria (DLCN-Criteria), Make Early Diagnosis to Prevent Early Deaths (MEDPED) criteria, and the Simon Broome Register Criteria--within national registries in order to define possible, probable, and definite cases of FH. The national registries used for this study are the Myocardial Ischaemia National Audit Project (MINAP) and National Audit of Percutaneous Coronary Intervention (BCIS) audit.

Following scoring of patients, a one-year and 30-day survival model were created in order to assess the effect of elevated cholesterol on survival, as suspected FH patients will have elevated cholesterol levels.

Data within MINAP ranges from 2003-2013 and data from BCIS ranges from 2007-2014.

Patient information within the audits was collected following admission to English and Welsh hospitals following a coronary event or percutaneous coronary intervention (PCI). Information related to survival and mortality was collected annually within each audit.

Participants for this study were those experiencing a premature cardiovascular event or coronary intervention (men <55 and women<60).

ELIGIBILITY:
Inclusion Criteria:

* Experienced a cardiac event and is therefore entered in CVD audit
* First registered event within audits

Exclusion Criteria:

* Under age 18
* Previous diagnosis of FH

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: UK based clinical population (participating hospitals across England and Wales).
Sampling Method: Non-Probability Sample
Enrollment: 1622948 (Actual)
Dates: Start 2003-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cholesterol (mmol/L) | Within 24 hours of Hospital Admission
  The primary outcome of this study is elevation of cholesterol due to suspected FH.
  Patients within either audit have experienced a major coronary event which is defined as: Myocardial Infarction (NSTEMI/STEMI), coronary artery bypass graft (CABG), aortic surgery, valve replacements/repairs, and percutaneous coronary intervention (PCI).
  This study is interested in detection of familial hypercholesterolaemia (FH) amongst patients experiencing a premature cardiac event. One of the key indicators of familial hypercholesterolaemia is elevated cholesterol.
  After hospital admission, a patient's cholesterol measurements will be taken within the first 24 hours. This is the only cholesterol measurement that is collected within the audit, as it does not fluctuate due to cholesterol depression post-event, and is potentially more indicative or a patient's cholesterol history (especially in situations where a patient has no prior history of statins).
Survival Following Hospital Admission for a Major Coronary Event | Up to 10 years
  Untreated familial hypercholesterolaemia--and as a result elevated cholesterol--may lead to premature death from coronary heart disease (CHD).
  Another primary outcome of this study is patient survival following hospital admission for a premature cardiac event.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Ayemoba, MSc, Study Chair — UCL; John Deanfield, MD, Principal Investigator — UCL; Owen Nicholas, PhD, Study Director — UCL; Riyaz Patel, MD, Study Chair — UCL

REFERENCES:
- [Background] Bell DA, Kirke AB, Barbour R, Southwell L, Pang J, Burrows S, Watts GF. Can patients be accurately assessed for familial hypercholesterolaemia in primary care? Heart Lung Circ. 2014 Dec;23(12):1153-7. doi: 10.1016/j.hlc.2014.06.015. Epub 2014 Jul 5. PMID 25065543
- [Background] Chen CX, Hay JW. Cost-effectiveness analysis of alternative screening and treatment strategies for heterozygous familial hypercholesterolemia in the United States. Int J Cardiol. 2015 Feb 15;181:417-24. doi: 10.1016/j.ijcard.2014.12.070. Epub 2014 Dec 24. PMID 25569270
- [Background] Futema M, Kumari M, Boustred C, Kivimaki M, Humphries SE. Would raising the total cholesterol diagnostic cut-off from 7.5 mmol/L to 9.3 mmol/L improve detection rate of patients with monogenic familial hypercholesterolaemia? Atherosclerosis. 2015 Apr;239(2):295-8. doi: 10.1016/j.atherosclerosis.2015.01.028. Epub 2015 Jan 28. PMID 25682026
- [Background] Goldberg AC, Hopkins PN, Toth PP, Ballantyne CM, Rader DJ, Robinson JG, Daniels SR, Gidding SS, de Ferranti SD, Ito MK, McGowan MP, Moriarty PM, Cromwell WC, Ross JL, Ziajka PE. Familial hypercholesterolemia: screening, diagnosis and management of pediatric and adult patients: clinical guidance from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Clin Lipidol. 2011 May-Jun;5(3):133-140. doi: 10.1016/j.jacl.2011.03.001. Epub 2011 Mar 11. PMID 21600517
- [Background] Gray J, Jaiyeola A, Whiting M, Modell M, Wierzbicki AS. Identifying patients with familial hypercholesterolaemia in primary care: an informatics-based approach in one primary care centre. Heart. 2008 Jun;94(6):754-8. doi: 10.1136/hrt.2006.107391. Epub 2007 Jun 17. PMID 17575326
- [Background] Haralambos K, Whatley SD, Edwards R, Gingell R, Townsend D, Ashfield-Watt P, Lansberg P, Datta DB, McDowell IF. Clinical experience of scoring criteria for Familial Hypercholesterolaemia (FH) genetic testing in Wales. Atherosclerosis. 2015 May;240(1):190-6. doi: 10.1016/j.atherosclerosis.2015.03.003. Epub 2015 Mar 6. PMID 25797312
- [Background] Kirke AB, Barbour RA, Burrows S, Bell DA, Vickery AW, Emery J, Watts GF. Systematic detection of familial hypercholesterolaemia in primary health care: a community based prospective study of three methods. Heart Lung Circ. 2015 Mar;24(3):250-6. doi: 10.1016/j.hlc.2014.09.011. Epub 2014 Sep 30. PMID 25445428
- [Background] Kirke A, Watts GF, Emery J. Detecting familial hypercholesterolaemia in general practice. Aust Fam Physician. 2012 Dec;41(12):965-8. PMID 23210121
- [Background] Nair DR, Sharifi M, Al-Rasadi K. Familial hypercholesterolaemia. Curr Opin Cardiol. 2014 Jul;29(4):381-8. doi: 10.1097/HCO.0000000000000083. PMID 24870549
- [Background] Nice.org.uk,. 'Identification And Management Of Familial Hypercholesterolaemia | Guidance And Guidelines | NICE'. N.p., 2008. Web. 27 Apr. 2015.
- [Background] Watts GF, Shaw JE, Pang J, Magliano DJ, Jennings GL, Carrington MJ. Prevalence and treatment of familial hypercholesterolaemia in Australian communities. Int J Cardiol. 2015 Apr 15;185:69-71. doi: 10.1016/j.ijcard.2015.03.027. Epub 2015 Mar 3. No abstract available. PMID 25791093
- [Background] Weng SF, Kai J, Andrew Neil H, Humphries SE, Qureshi N. Improving identification of familial hypercholesterolaemia in primary care: derivation and validation of the familial hypercholesterolaemia case ascertainment tool (FAMCAT). Atherosclerosis. 2015 Feb;238(2):336-43. doi: 10.1016/j.atherosclerosis.2014.12.034. Epub 2014 Dec 20. PMID 25555265
- [Background] Arnold SV, Kosiborod M, Tang F, Zhao Z, McCollam PL, Birt J, Spertus JA. Changes in low-density lipoprotein cholesterol levels after discharge for acute myocardial infarction in a real-world patient population. Am J Epidemiol. 2014 Jun 1;179(11):1293-300. doi: 10.1093/aje/kwu060. Epub 2014 Apr 16. PMID 24743066
- [Background] Austin MA, Hutter CM, Zimmern RL, Humphries SE. Genetic causes of monogenic heterozygous familial hypercholesterolemia: a HuGE prevalence review. Am J Epidemiol. 2004 Sep 1;160(5):407-20. doi: 10.1093/aje/kwh236. PMID 15321837
- [Background] Barth JH, Jackson BM, Farrin AJ, Efthymiou M, Worthy G, Copeland J, Bailey KM, Romaine SP, Balmforth AJ, McCormack T, Whitehead A, Flather MD, Nixon J, Hall AS; SPACE ROCKET Trial Group. Change in serum lipids after acute coronary syndromes: secondary analysis of SPACE ROCKET study data and a comparative literature review. Clin Chem. 2010 Oct;56(10):1592-8. doi: 10.1373/clinchem.2010.145631. Epub 2010 Aug 20. PMID 20729301
- [Background] Besseling J, Kindt I, Hof M, Kastelein JJ, Hutten BA, Hovingh GK. Severe heterozygous familial hypercholesterolemia and risk for cardiovascular disease: a study of a cohort of 14,000 mutation carriers. Atherosclerosis. 2014 Mar;233(1):219-23. doi: 10.1016/j.atherosclerosis.2013.12.020. Epub 2014 Jan 11. PMID 24529147
- [Background] Chakko S, Myerburg RJ. Cardiac complications of cocaine abuse. Clin Cardiol. 1995 Feb;18(2):67-72. doi: 10.1002/clc.4960180206. PMID 7720292
- [Background] Charniak, Eugene. 'Bayesian Networks Without Tears'. AI Magazine 12.4 (1991): 50-63. Print.
- [Background] De Castro-Orós, Isabel, Miguel Pocoví, and Fernando Civeira. 'The Fine Line Between Familial And Polygenic Hypercholesterolemia'. Clinical Lipidology 8.3 (2013): 303-306. Web.
- [Background] de Ferranti SD, de Boer IH, Fonseca V, Fox CS, Golden SH, Lavie CJ, Magge SN, Marx N, McGuire DK, Orchard TJ, Zinman B, Eckel RH. Type 1 diabetes mellitus and cardiovascular disease: a scientific statement from the American Heart Association and American Diabetes Association. Circulation. 2014 Sep 23;130(13):1110-30. doi: 10.1161/CIR.0000000000000034. Epub 2014 Aug 11. No abstract available. PMID 25114208
- [Background] Gaziano JM, Hennekens CH, Satterfield S, Roy C, Sesso HD, Breslow JL, Buring JE. Clinical utility of lipid and lipoprotein levels during hospitalization for acute myocardial infarction. Vasc Med. 1999;4(4):227-31. doi: 10.1177/1358836X9900400404. PMID 10613626
- [Background] Kasim S, O'Donabhain R, Mcfadden E. Cocaine-associated myocardial infarction: should they all be stented? Case Rep Cardiol. 2011;2011:347806. doi: 10.1155/2011/347806. Epub 2011 Jul 19. PMID 24826216
- [Background] Mabuchi H, Higashikata T, Nohara A, Lu H, Yu WX, Nozue T, Noji Y, Katsuda S, Kawashiri MA, Inazu A, Kobayashi J, Koizumi J. Cutoff point separating affected and unaffected familial hypercholesterolemic patients validated by LDL-receptor gene mutants. J Atheroscler Thromb. 2005;12(1):35-40. doi: 10.5551/jat.12.35. PMID 15725694
- [Background] Mittleman MA, Mintzer D, Maclure M, Tofler GH, Sherwood JB, Muller JE. Triggering of myocardial infarction by cocaine. Circulation. 1999 Jun 1;99(21):2737-41. doi: 10.1161/01.cir.99.21.2737. PMID 10351966
- [Background] Mundal L, Sarancic M, Ose L, Iversen PO, Borgan JK, Veierod MB, Leren TP, Retterstol K. Mortality among patients with familial hypercholesterolemia: a registry-based study in Norway, 1992-2010. J Am Heart Assoc. 2014 Dec 2;3(6):e001236. doi: 10.1161/JAHA.114.001236. PMID 25468658
- [Background] Nordestgaard BG, Chapman MJ, Humphries SE, Ginsberg HN, Masana L, Descamps OS, Wiklund O, Hegele RA, Raal FJ, Defesche JC, Wiegman A, Santos RD, Watts GF, Parhofer KG, Hovingh GK, Kovanen PT, Boileau C, Averna M, Boren J, Bruckert E, Catapano AL, Kuivenhoven JA, Pajukanta P, Ray K, Stalenhoef AF, Stroes E, Taskinen MR, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia is underdiagnosed and undertreated in the general population: guidance for clinicians to prevent coronary heart disease: consensus statement of the European Atherosclerosis Society. Eur Heart J. 2013 Dec;34(45):3478-90a. doi: 10.1093/eurheartj/eht273. Epub 2013 Aug 15. PMID 23956253
- [Background] Orchard TJ, Costacou T, Kretowski A, Nesto RW. Type 1 diabetes and coronary artery disease. Diabetes Care. 2006 Nov;29(11):2528-38. doi: 10.2337/dc06-1161. No abstract available. PMID 17065698
- [Background] Qureshi AI, Chaudhry SA, Suri MF. Cocaine use and the likelihood of cardiovascular and all-cause mortality: data from the Third National Health and Nutrition Examination Survey Mortality Follow-up Study. J Vasc Interv Neurol. 2014 May;7(1):76-82. PMID 24920992
- [Background] Raal FJ, Pilcher GJ, Panz VR, van Deventer HE, Brice BC, Blom DJ, Marais AD. Reduction in mortality in subjects with homozygous familial hypercholesterolemia associated with advances in lipid-lowering therapy. Circulation. 2011 Nov 15;124(20):2202-7. doi: 10.1161/CIRCULATIONAHA.111.042523. Epub 2011 Oct 10. PMID 21986285
- [Background] Schnell O, Cappuccio F, Genovese S, Standl E, Valensi P, Ceriello A. Type 1 diabetes and cardiovascular disease. Cardiovasc Diabetol. 2013 Oct 28;12:156. doi: 10.1186/1475-2840-12-156. PMID 24165454
- [Background] Sijbrands EJ, Westendorp RG, Defesche JC, de Meier PH, Smelt AH, Kastelein JJ. Mortality over two centuries in large pedigree with familial hypercholesterolaemia: family tree mortality study. BMJ. 2001 Apr 28;322(7293):1019-23. doi: 10.1136/bmj.322.7293.1019. PMID 11325764
- [Background] Spiegelhalter, D. J, K. R Abrams, and Jonathan P Myles. Bayesian Approaches To Clinical Trials And Health-Care Evaluation. Chichester: John Wiley & Sons, 2004. Print.
- [Background] Stein EA, Raal FJ. Polygenic familial hypercholesterolaemia: does it matter? Lancet. 2013 Apr 13;381(9874):1255-7. doi: 10.1016/S0140-6736(13)60187-7. Epub 2013 Feb 22. No abstract available. PMID 23433574
- [Background] Sterne JA, White IR, Carlin JB, Spratt M, Royston P, Kenward MG, Wood AM, Carpenter JR. Multiple imputation for missing data in epidemiological and clinical research: potential and pitfalls. BMJ. 2009 Jun 29;338:b2393. doi: 10.1136/bmj.b2393. PMID 19564179
- [Background] Versmissen J, Oosterveer DM, Yazdanpanah M, Defesche JC, Basart DC, Liem AH, Heeringa J, Witteman JC, Lansberg PJ, Kastelein JJ, Sijbrands EJ. Efficacy of statins in familial hypercholesterolaemia: a long term cohort study. BMJ. 2008 Nov 11;337:a2423. doi: 10.1136/bmj.a2423. PMID 19001495
- [Background] Wald DS, Bangash FA, Bestwick JP. Prevalence of DNA-confirmed familial hypercholesterolaemia in young patients with myocardial infarction. Eur J Intern Med. 2015 Mar;26(2):127-30. doi: 10.1016/j.ejim.2015.01.014. Epub 2015 Feb 11. PMID 25682442
- [Background] Wattanasuwan N, Khan IA, Gowda RM, Vasavada BC, Sacchi TJ. Effect of acute myocardial infarction on cholesterol ratios. Chest. 2001 Oct;120(4):1196-9. doi: 10.1378/chest.120.4.1196. PMID 11591560
- [Background] World Health Organization,. Familial Hypercholesterolaemia. Geneva, Switzerland: Human Genetics Programme, 1998. Print. Annex Progress Report.
- [Background] Sun LY, Zhang YB, Jiang L, Wan N, Wu WF, Pan XD, Yu J, Zhang F, Wang LY. Erratum: Identification of the gene defect responsible for severe hypercholesterolaemia using whole-exome sequencing. Sci Rep. 2015 Aug 3;5:12656. doi: 10.1038/srep12656. No abstract available. PMID 26237740
- [Background] Mortality in treated heterozygous familial hypercholesterolaemia: implications for clinical management. Scientific Steering Committee on behalf of the Simon Broome Register Group. Atherosclerosis. 1999 Jan;142(1):105-12. PMID 9920511
- [Background] Moons KG, Donders RA, Stijnen T, Harrell FE Jr. Using the outcome for imputation of missing predictor values was preferred. J Clin Epidemiol. 2006 Oct;59(10):1092-101. doi: 10.1016/j.jclinepi.2006.01.009. Epub 2006 Jun 19. PMID 16980150
- [Background] Medeiros AM, Alves AC, Bourbon M. Mutational analysis of a cohort with clinical diagnosis of familial hypercholesterolemia: considerations for genetic diagnosis improvement. Genet Med. 2016 Apr;18(4):316-24. doi: 10.1038/gim.2015.71. Epub 2015 May 28. PMID 26020417
- [Background] McAllister KS, Ludman PF, Hulme W, de Belder MA, Stables R, Chowdhary S, Mamas MA, Sperrin M, Buchan IE; British Cardiovascular Intervention Society and the National Institute for Cardiovascular Outcomes Research. A contemporary risk model for predicting 30-day mortality following percutaneous coronary intervention in England and Wales. Int J Cardiol. 2016 May 1;210:125-32. doi: 10.1016/j.ijcard.2016.02.085. Epub 2016 Feb 17. PMID 26942330
- [Background] Marks D, Thorogood M, Neil HA, Humphries SE. A review on the diagnosis, natural history, and treatment of familial hypercholesterolaemia. Atherosclerosis. 2003 May;168(1):1-14. doi: 10.1016/s0021-9150(02)00330-1. PMID 12732381
- [Background] Do R, Stitziel NO, Won HH, Jorgensen AB, Duga S, Angelica Merlini P, Kiezun A, Farrall M, Goel A, Zuk O, Guella I, Asselta R, Lange LA, Peloso GM, Auer PL; NHLBI Exome Sequencing Project; Girelli D, Martinelli N, Farlow DN, DePristo MA, Roberts R, Stewart AF, Saleheen D, Danesh J, Epstein SE, Sivapalaratnam S, Hovingh GK, Kastelein JJ, Samani NJ, Schunkert H, Erdmann J, Shah SH, Kraus WE, Davies R, Nikpay M, Johansen CT, Wang J, Hegele RA, Hechter E, Marz W, Kleber ME, Huang J, Johnson AD, Li M, Burke GL, Gross M, Liu Y, Assimes TL, Heiss G, Lange EM, Folsom AR, Taylor HA, Olivieri O, Hamsten A, Clarke R, Reilly DF, Yin W, Rivas MA, Donnelly P, Rossouw JE, Psaty BM, Herrington DM, Wilson JG, Rich SS, Bamshad MJ, Tracy RP, Cupples LA, Rader DJ, Reilly MP, Spertus JA, Cresci S, Hartiala J, Tang WH, Hazen SL, Allayee H, Reiner AP, Carlson CS, Kooperberg C, Jackson RD, Boerwinkle E, Lander ES, Schwartz SM, Siscovick DS, McPherson R, Tybjaerg-Hansen A, Abecasis GR, Watkins H, Nickerson DA, Ardissino D, Sunyaev SR, O'Donnell CJ, Altshuler D, Gabriel S, Kathiresan S. Exome sequencing identifies rare LDLR and APOA5 alleles conferring risk for myocardial infarction. Nature. 2015 Feb 5;518(7537):102-6. doi: 10.1038/nature13917. Epub 2014 Dec 10. PMID 25487149
- [Background] Damgaard D, Larsen ML, Nissen PH, Jensen JM, Jensen HK, Soerensen VR, Jensen LG, Faergeman O. The relationship of molecular genetic to clinical diagnosis of familial hypercholesterolemia in a Danish population. Atherosclerosis. 2005 May;180(1):155-60. doi: 10.1016/j.atherosclerosis.2004.12.001. Epub 2005 Jan 12. PMID 15823288
- [Background] Civeira F, Ros E, Jarauta E, Plana N, Zambon D, Puzo J, Martinez de Esteban JP, Ferrando J, Zabala S, Almagro F, Gimeno JA, Masana L, Pocovi M. Comparison of genetic versus clinical diagnosis in familial hypercholesterolemia. Am J Cardiol. 2008 Nov 1;102(9):1187-93, 1193.e1. doi: 10.1016/j.amjcard.2008.06.056. Epub 2008 Aug 27. PMID 18940289
- [Background] Benn M, Watts GF, Tybjaerg-Hansen A, Nordestgaard BG. Familial hypercholesterolemia in the danish general population: prevalence, coronary artery disease, and cholesterol-lowering medication. J Clin Endocrinol Metab. 2012 Nov;97(11):3956-64. doi: 10.1210/jc.2012-1563. Epub 2012 Aug 14. PMID 22893714
- [Background] Al-Rasadi K, Al-Waili K, Al-Sabti HA, Al-Hinai A, Al-Hashmi K, Al-Zakwani I, Banerjee Y. Criteria for Diagnosis of Familial Hypercholesterolemia: A Comprehensive Analysis of the Different Guidelines, Appraising their Suitability in the Omani Arab Population. Oman Med J. 2014 Mar;29(2):85-91. doi: 10.5001/omj.2014.22. PMID 24715932
- [Background] Cattle BA, Baxter PD, Greenwood DC, Gale CP, West RM. Multiple imputation for completion of a national clinical audit dataset. Stat Med. 2011 Sep 30;30(22):2736-53. doi: 10.1002/sim.4314. Epub 2011 Jul 22. PMID 21786284